CLINICAL TRIAL: NCT01314274
Title: A Randomized Double Blind Placebo Controlled Trial of Intranasal Submucosal Bevacizumab in Hereditary Hemorrhagic Telangiectasia
Brief Title: Intranasal Submucosal Bevacizumab for Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Martin Burian, Prof. Dr. Martin Burian, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: bevacizumab HHT; 2009-018049-19 (EudraCT Number)
Record Dates: First submitted 2011-03-09; First posted 2011-03-14 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: HHT; Morbus Osler; Epistaxis
Keywords: Epistaxis; Osler; Weber; Rendu; HHT; Hereditary haemorrhagic telangiectasia
MeSH Terms: conditions — Epistaxis; Telangiectasia, Hereditary Hemorrhagic | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- bevacizumab (Experimental): submucosal intranasal bevacizumab on day 0
  Interventions: Drug: Bevacizumab
- placebo (Placebo Comparator): 0.9% NaCl intranasal submucosal on day 0
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Bevacizumab — 100mg intranasal submucosal bevacizumab in 10ml
  Arms: bevacizumab
Drug: NaCl — 10ml of 0.9% NaCl intranasal submucosal
  Arms: placebo

SUMMARY:
In a case series intranasal submucosal bevacizumab has been shown to reduce epistaxis in patients suffering from Hereditary Haemorrhagic Telangiectasia together with KTP Laser therapy. The aim of this study is to evaluate the effectiveness of submucosal intranasal bevacizumab compared to placebo in a randomized double blind trial setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and staged HHT (Shovlin et al 2000)
* Age 18-80
* Minimum of 2 episodes of epistaxis/ week
* Ability and willingness to complete diary and comply with study requirements.

Exclusion Criteria:

* Uncontrolled hypertension (systolic blood pressure > 150mmHg, diastolic blood pressure > 90mmHg)
* History of a thromboembolic event, including myocardial infarction or cerebral vascular accident
* Malignancy of the upper respiratory tract within the last year
* Recent (<3 months) or planned surgery
* Proteinuria
* Nasal intervention (Laser or Cautery) in pretreatment phase
* Allergy to local anesthetic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
relative change in average daily Epistaxis VAS scores compared to baseline | day 10 - 84 posttreatment
  Daily epistaxis VAS scores are recorded in a diary. The baseline score is the average daily epistaxis VAS score 4 weeks before treatment (day -28 to 0). This score is compared to the average daily VAS score day 10-84 posttreatment. The relative change of this average score compared to baseline is the primary outcome.

SECONDARY OUTCOMES:
Epistaxis Severity Score HHT-ESS compared to baseline | 3 months post treatment
Epistaxis frequency, duration and severity compared to baseline | day 10 - 84 posttreatment
Number of emergency department visits due to epistaxis compared to baseline | day 10 - 84 posttreatment
lab results (ferritin values, Hb, Hct) compared to baseline | day 84 posttreatment
Number of transfusions needed compared to baseline | day 10-84 posttreatment
Average daily epistaxis VAS scores compared to baseline among age groups and among groups with different epistaxis severity | day 10-84 posttreatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik für HNO, Medizinische Univeristät Wien, Vienna, Austria

REFERENCES:
- [Derived] Riss D, Burian M, Wolf A, Kranebitter V, Kaider A, Arnoldner C. Intranasal submucosal bevacizumab for epistaxis in hereditary hemorrhagic telangiectasia: a double-blind, randomized, placebo-controlled trial. Head Neck. 2015 Jun;37(6):783-7. doi: 10.1002/hed.23655. Epub 2014 Apr 30. PMID 24595923